CLINICAL TRIAL: NCT04160429
Title: Pilot Study to Evaluate Substances in Sweat, Saliva, and Blood
Brief Title: Biospecimen Analysis in Detecting Chemical Concentrations in Patients With Chronic or Infectious Diseases Receiving Meditations
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18380; NCI-2019-07380 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18380 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Chronic Disease; Infectious Disorder
MeSH Terms: conditions — Chronic Disease; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sweat, saliva, and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Device feasibility (Macroduct Sweat Collection System): Patients undergo collection of sweat samples via Macroduct Sweat Collection System 3710S and saliva and blood samples within 24 hours after medication administrations. Patients also complete questionnaires over 5-10 minutes and have medical charts reviewed.
  Interventions: Procedure: Biospecimen Collection; Other: Medical Chart Review; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of sweat, saliva, and blood samples
Other: Medical Chart Review — Review of medical chart
  Other Names: Chart Review
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This trial collects and analyzes sweat and saliva samples compared to blood in detecting chemical concentrations in the body in patients with chronic or infectious diseases receiving medications. Wearable sweat sensors are capable of monitoring electrolytes and metabolites (sodium, potassium, glucose, lactate, etc.) for health monitoring and disease diagnosis. Designing wearable sweat sensors capable of providing information regarding drug administration may be challenging due to ultralow concentrations in biofluids. This trial seeks to determine if the use of a smart wristband can accurately measure the levels of chemicals and substances in sweat.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare novel, home-based methods of quantitating medication concentrations in either saliva or sweat to the 'gold standard' of liquid chromatography - mass spectrometry of plasma.

SECONDARY OBJECTIVES:

I. To compare novel home-based methods of quantitating substances in either saliva or sweat to the 'gold standard' in plasma.

II. Assess the ease of obtaining home-based samples.

OUTLINE:

Patients undergo collection of sweat samples via Macroduct Sweat Collection System 3710S and saliva and blood samples within 24 hours after medication administrations. Patients also complete questionnaires over 5-10 minutes and have medical charts reviewed.

After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to receive medications including, but not limited to, cyclophosphamide, mycophenolic acid, mycophenolate mofetil, metformin or busulfan (any dose, any number of doses, any dosing frequency) as part of treatment at any time. Patients with chronic or infectious diseases can participate
* Willingness to:

  * Provide blood, sweat, and saliva samples
  * Permit medical record review

Exclusion Criteria:

* Pilocarpine allergy
* Difficulty with understanding written English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic or infectious diseases scheduled to receive medications
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2029-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Predictive performance of the home-based sampling | Up to 4 hours
  Will be assessed by Pearson correlation and quantification of the predictive performance. The predictive performance of the home-based sampling methods will be assessed by calculating the median percentage prediction error (MPPE).
Observed plasma concentrations | Up to 4 hours
  Will be assessed by Pearson correlation and quantification of the predictive performance. The values from plasma will be considered the observed concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannine S McCune, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States